CLINICAL TRIAL: NCT05537415
Title: Prevalence of Medical Care in an Emergency Structure and Expectations Vis-à-vis the Care System Among Women Victims of Violence Within the Couple Treated in the Associative, Social and Medico-legal Environment
Brief Title: Prevalence of Medical Care in an Emergency Structure of the Women Victims of Violence Within the Couple
Acronym: Spousal-Abuse
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8698
Record Dates: First submitted 2022-09-09; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Spousal-Abuse
Keywords: Spousal-Abuse; Violence against women

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Violence against women within the couple is a major socio-political and public health problem.

Indeed, in 2020, 219,000 women were victims of violence within their couple and 102 women were killed by their partner or ex-partner.

On average, the number of women aged 18 to 75 who in the course of a year are victims of rape and/or attempted rape is estimated at 94,000 women, and in 47% of cases it is the spouse or the ex-spouse who is the author of the facts.

This violence has major health and social consequences: the leading cause of death and disability among women aged 16 to 44 in Europe. In France, a woman dies as a result of domestic violence every 2.5 days and the overall cost of domestic violence in 2012 amounted to 3.6 billion euros in France.

A better knowledge of the use of care for wives of victims of violence and their feelings vis-à-vis the medical care in an emergency service will make it possible to identify the problems related to their care based on their feelings. of these patients, to understand why they would not have consulted as a first resort if necessary and to subsequently propose avenues for improvement.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (age ≥ 18 years old)
* victims of violence committed within the couple
* Initial visit to the emergency room or not
* Subject not opposed to participating in the study

Exclusion Criteria:

* Intra-family violence committed by a parent, outside the couple (for example: father, grandfather, brother, cousin, uncle, child)
* Impossibility of giving informed information to the subject (subject in an emergency situation, difficulties in understanding the subject, etc.)

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Adult women (age ≥ 18 years old) victims of violence committed within the couple
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of recourse to care in an emergency structure among women cared for in a reception center for women victims of violence | from January 01, 2012 to December 31, 2022

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'accueil des urgences - CHU de Strasbourg - France, Strasbourg, France